# Pharmacogenomics of the Variability in the *In Vivo* Response to Glucocorticoids

NCT03023891

10/23/17

**Vivian K. Kawai, M.D.**Division of Clinical Pharmacology

# **Table of Contents:**

# **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Animal Studies and Previous Human Studies
- 4.0 Inclusion/Exclusion Criteria
- 5.0 Enrollment/Randomization
- **6.0 Study Procedures**
- 7.0 Risks of Investigational Agents/Devices (side effects)
- 8.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 9.0 Study Withdrawal/Discontinuation
- **10.0 Statistical Considerations**
- 11.0 Privacy/Confidentiality Issues
- 12.0 Follow-up and Record Retention

# 1.0 Background

Glucocorticoids (GCs) are commonly used worldwide to treat several conditions, including asthma, lymphomas, and chronic inflammatory disorders.  $^{1.2}$  It is estimated that between 1-3% of the general population in developed countries have used GCs, and that 65-75% of these patients used GCs chronically ( $\geq$  3 months).  $^{1.3}$  Although GCs have dramatic anti-inflammatory and immunosuppressive effects, they exhibit **large interindividual variability in GC response in terms of efficacy and toxicity**. This variability in GC response explains why nearly 30% of patients with different pathological conditions have a suboptimal response to the anti-inflammatory effects of GCs<sup>4-7</sup> resulting in morbidity and substantial economic costs. Moreover, it explains why between 10 to 80% of patients who receive GCs chronically develop serious side effects.  $^{9-11}$ 

# 2.0 Rationale and Specific Aims

The large inter-individual variability in GC response has a genetic component, but the genetic architecture of GC response is still unknown. A few studies have linked a small number of genetic variants with GC therapeutic efficacy. 12-15 One reason for the lack of progress in identifying the genetic determinants of GC efficacy has been the measurement of response in clinically heterogeneous phenotypes (e.g., asthma, inflammatory bowel disease). These phenotypes require weeks to respond to GCs, and the pharmacogenetic signal is susceptible to confounding by disease heterogeneity and co-therapies. A more attractive approach is to study a "clean" intermediate phenotype — a pharmacodynamic measure of GC efficacy. GC-induced lymphopenia is such a measure; this is a rapid, reproducible, dose- and concentration-dependent response that has been quantified in human pharmacokinetic and pharmacodynamic models. 16-19 Moreover, lymphocytes are major determinants of inflammation and GCs exert part of their anti-inflammatory effects by altering lymphocyte kinetics and survival. Thus, GC-induced lymphopenia is a robust and relevant intermediate phenotype to study the genetic predictors of GC efficacy.

In addition to variability in GC efficacy, there is also marked variability in the frequency and severity of GC toxicity. One of the most common metabolic side effects of GC therapy is GC-induced glucose intolerance. Although GC impairs glucose metabolism through insulin resistance and by  $\beta$ -cell dysfunction, there is large variability in the severity of the metabolic effects of GCs that is explained by clinical factors. Evidence suggest that metabolic effects of GC has a genetic component, but the genetic determinants of metabolic toxicity remains unknown.

As other complex traits, genome-wide association studies (GWAS) have identified some risk variants for GC response; 12-15 however the functional relevance for most of these variants are not known. In complex traits, the combination of GWAS information and large gene expression data has shown that top hits on GWAS were enriched for polymorphisms that regulate expression levels of genes (regulatory polymorphisms), 23 and that these regulatory variants explained a large proportion of the phenotypic variability for complex phenotypes including drug response. 24, 25

GCs are known to exert their effect through changes in gene expression and also by interacting with several transcription factors, <sup>26,27</sup> but we still do not know which genes are involved in the response to *in vivo* administration GC in humans, and which genetic variants are more likely to affect the expression of these genes. Thus, we propose to perform a hypothesis-generating pilot study to identify potential set of genes and

regulatory variants that are likely to be involve in the response to GC in terms of efficacy and metabolic toxicity.

For this pilot study we plan to use a robust pharmacodynamic effect of GCs (GC-induced lymphopenia) and a common metabolic complication of GC therapy (GC-induced glucose intolerance) after *in vivo* administration of GC as our clinical phenotypes to:

**Specific Aim:** To characterize gene expression patterns that are predictive of *in vivo* GC response, and identify regulatory variants that are associated with *in vivo* GC response by challenging 40 healthy volunteers with 60 mg of oral prednisone. We will measure changes in lymphocyte counts and changes in glucose regulation (using the 75 gr glucose tolerance test ~ OGTT) as surrogates of GC efficacy and metabolic toxicity. We will perform transcriptome-wide next generation RNA sequencing to measure changes in gene expression due to *in vivo* administration of GC and study the association of gene expression patterns with our clinical phenotypes. Once we identify a set of genes that are significantly changed after *in vivo* GC administration, we will select potential regulatory variants that have been associated with changes in expression of these genes in public available expression quantitative trait loci (eQTL) datasets to perform genome interrogation and eQTL analysis. This will allow us to identify variants that are associated with gene expression changes due to *in vivo* administration of GC.

#### 3.0 Animal Studies and Previous Human Studies

Pharmacodynamic measures of GC efficacy: One of the mechanism through which GC exerts its anti-inflammatory effects is by modifying the traffic and function of immune cells. 18,28,29 GCs markedly increase the number of circulating neutrophils and decrease the number of circulating white blood cells (WBC). 40,30,31 Among WBC, neutrophils and lymphocytes have been largely use to study the pharmacodynamics of GCs; 16,17,32,33 mostly because the other leukocytes represent a small percentage of the circulating WBC and the administration of GCs reduced greatly their number (sometimes to undetectable levels) making difficult to establish a dose-concentration response. 14 Not only the changes induced by GCs in circulating neutrophil and lymphocyte counts are dose- and concentration-dependent, 14 reproducible, 15 and obtained with equivalent doses of commonly used GCs; 16 but also the same response can be evoked in healthy individuals and in patients with inflammatory disorders. 14,36,37 Thus, changes in WBC counts are well-established and reproducible pharmacodynamic phenotypes to study the genetics of GC response.

**Metabolic side effects of GCs – glucose intolerance**: There is also large variability in GC toxicity. Glucose intolerance is a frequent and clinically relevant metabolic complication of GC therapy<sup>21,22</sup> that can lead to transient hyperglycemia<sup>38</sup> or to a permanent condition called GC-induced diabetes.<sup>39,40</sup> The mechanisms through which GCs induce glucose intolerance are similar to those involved in the development of type 2 diabetes mellitus (T2DM),<sup>39,41,42</sup> and include insulin resistance<sup>43</sup> and β-cell dysfunction.<sup>44,45</sup> Hyperglycemia occurs when β-cell failure can no longer compensate for the degree of insulin resistance. Clinical studies have shown that short-term administration of GCs impairs glucose tolerance in individuals with normal glucose tolerance;<sup>44,46,48</sup> while a high single doses of GCs have shown to increase insulin resistance<sup>44,46,48,49</sup> and consequently increase insulin secretion<sup>44,46</sup> a compensatory mechanism that is reduced in individuals at risk for T2DM.<sup>44,48,50-53</sup> Evidence suggest that

glucose intolerance during GC therapy is in part due to a genetic component since the degree of glucose intolerance varies markedly among patients who received the same dose of GCs;<sup>54</sup> there is large variability in the incidence of glucose intolerance due to GC therapy among races;<sup>55,56</sup> and variants known to affect GC sensitivity have been associated with metabolic phenotypes<sup>57-65</sup> Despite these observations, the genetic determinants of GC–induce metabolic toxicity are not known and we cannot predict who will develop a metabolic complication during GC therapy.

GC exert their effects through the regulation of gene expression by regulatory variants: GCs are known to exert their effect through changes in gene expression and by interacting with several transcription factors. Thus, they represent an excellent tool to study gene-environment interactions.66 Accordingly, using immortalized and cultured human peripheral blood mononuclear cells (PBMCs), several studies have shown that GC response is associated with different patterns of transcriptional response, 14,27,67 and that variants in regulatory binding sites at GC-targeted genes may play a role in GC response variabilty. 12,14,26,27 However, the process of immortalization and the culture of cells are known to affect the gene expression response and likely differ from in vivo expression. 68-70 Moreover, the eQTL studies using immortalized cells have little overlap with eQTL from cultured cells.<sup>27</sup> To our knowledge, there is only one small study that has examine gene expression changes with in vivo administration with GC but have not performed eQTL analysis. Olnes explored genome transcription response after in vivo administration of GCs using whole transcriptome microarrays, 71 and found that peak changes in gene expression were observed 4 hours after GC administration with large variability in the gene expression changes. We propose to extend Olnes' work by studying the role that genetic variants have in the observed variability of gene expression response during in vivo administration of GC. Besides, we propose to study PBMCs gene expression response to a glucose challenge due to in vivo administration of GCs to study the genetic architecture of the metabolic complications of GC administration, which has not be done.

#### 4.0 Inclusion/Exclusion Criteria

#### Inclusion criteria:

- 18 to 45 years old (to exclude the effect of age on glucose tolerance)
- BMI between 20 and 30 kg/m² (to exclude individuals that are likely to have impaired insulin response)
- Normal fasting glucose
- Stable weight for three months before participation

#### Exclusion criteria:

- BMI ≥30kg/m²
- Fasting glucose ≥126 mg/dl
- Shift work or disordered sleep (to exclude individuals with alterations in the hypothalamus-adrenergic axis)
- Any active diseases (requiring current treatment)
- Use of any medication regularly (including over-the-counter such as aspirin, ibuprofen, etc)
- Previous exposure to GCs (within the last year)
- Diabetes
- Pregnant or breastfeeding

# 5.0 Enrollment/Randomization

We plan to recruit participants by sending notices through ResearchMatch.org, Research notifications email, word of mouth, and fliers.

# **6.0 Study Procedures**

Potential participants will meet with the study team to discuss the purpose, inclusion and exclusion criteria, procedures and risk/benefits of the study. Those who sign the consent form will come for a screening visit, and if they fulfill inclusion and exclusion criteria, they will come to Vanderbilt University Medical Center (VUMC) for two study visits in the following 30 days. The study visits will take place within a one-month window, will start early in the morning and will last approximately 6 hours. For all the study visits participants will be asked to fast overnight and avoid alcohol consumption and exercise (except walking<30 minutes) 48 hours before the visit, and be free of any illness.

- Screening visit: The participant will arrive fasting early in the morning to VUMC. In this visit, the study team will ask questions about his/her health and past medical history. The study team will perform a brief physical exam that include participant's height and weight to calculate the body mass index (BMI) and waist and hip circumference. Blood samples will be collected for safety reasons and to culture peripheral blood mononuclear cells *in vitro* with glucocorticoid. We will request a urine and stool sample for future research. Women of child-bearing potential will have a urine pregnancy test. Women who are pregnant will not be allowed to participate. The study team will provide instructions about fasting and activities before the study visits. If any of the test results on the blood collected at the screening suggests that the participant may have a condition that can alter the study (e.g., random glucose>200 mg/dL) or put him/her at risk, the study team will contact the participant to explain the reason why he/she cannot participate in the study.
- Study visit 1: The participant will arrive fasting early in the morning to VUMC. A standardized clinical interview and brief physical examination will be performed. For female participants, a urine sample will be collected for pregnancy testing. A fingerstick will be perform to check fasting glucose level. An intravenous catheter will be placed in one arm for continuous sampling around 31/2 hours after the participant arrival. Once venous access is secure, blood samples will be collected at different times. If the fasting glucose is ≥126 mg/dl, the participant will be excluded from the oral glucose tolerance test study, and blood will be collected approximately 4 and 6 hours after the fingerstick. If blood glucose is below 126 mg/dl; we will collect blood samples around 4 hours after the patient's arrival. Immediately afterwards, a 75-gram glucose solution will be administered as part of the oral glucose tolerance test (OGTT), and blood samples will be collected at 10, 20, 30, 60, 90, and 120 minutes after glucose ingestion. Participants with 2-hour blood glucose ≥200mg/dl will be excluded. A standard meal will be provided at the end of the study visit.
- Study visit 2: Visit 2 will occur within one month after visit 1. An interview, physical exam, and urine testing in the fasting participant will be performed, as in Study visit 1. A single dose of 60 mg of oral prednisone will be administered immediately after a fingerstick for blood glucose is performed. Approximately 31/2 hours later, an intravenous catheter will be placed in one arm for continuous sampling. The first blood

collection will be perform around 4 hours after the ingestion of prednisone, and immediately after an OGTT will be performed (if tolerated on study visit 1). Blood collection will occur at 10, 20, 30, 60, 90, and 120 minutes after glucose ingestion. A standard meal will be provided at the end of the study visit.

Each visit will take approximately 6 hours and the participant should stay at VUMC during the study visits. The study team will contact the participant by phone for the next two consecutive days after the last visit to inquire about any problem related to the study.

Measurements: Blood samples will be used for the following:

- Basic metabolic screening
- Glucose, insulin, and C-peptide to study insulin sensitivity and  $\beta$  cell function<sup>72, 73</sup> at both study visits.
- Blood cell counts.
- RNA extraction will be performed from PBMCs collected in both study visits.
- Genotyping
- Urine and stool samples will be stored for future research. Female participants will have a urine pregnancy test at each study visit.

RNA sequence and Genotyping: RNA will be extracted from PBMC lysates following standard procedures and send to the Vanderbilt Technologies for Advance Genomics (VANTAGE) Core for RNA-seq. VANTAGE will perform RNA sequencing including small RNAs. Once sequencing data is available, VANGARD will align the reads to a reference genome, count the reads, compared gene expression levels before and after GC exposure and obtain a list of genes that are differential expressed. Genotyping will be performed at the VANTAGE Core using Megachip

#### 7.0 Risks

Drawing of venous blood: Puncturing of a vein may result in minor bleeding or bruising. Because some people may faint during blood draw, we will ask the participants to lie down during blood collection.

Fasting: Dizziness, light-headedness, or nausea can occur as result of fasting.

75gr OGTT: nausea, vomiting, or light-headedness may occur after drinking the glucose solution. A drop in blood glucose levels may occur during the test which may cause nausea, dizziness, sweating, weakness, or restlessness. A significant drop in glucose levels during the test is likely to occur during illnesses, alcohol consumption, dieting, in patients using medications or long periods of bed rest (hospitalized patients), but rarely in healthy people. The study team will monitor the blood glucose several times during the test using a glucometer. If blood glucose levels fall out of safe ranges, the test will be stopped and oral (or intravenous) glucose solutions will be administered if needed. Transient hyperglycemia during OGTT is likely to occur in people with undiagnosed diabetes, and it resolves spontaneously once the test is complete.

Prednisone is a FDA-approved drug for several disorders. Glucocorticoids have several side effects (e.g., increase in blood pressure, electrolytes abnormalities, adrenocortical suppression, risk of infection, mood and behavioral disturbance, gastrointestinal problems, etc.), which are more likely to occur with repeated and high doses. We plan to administer a single dose of prednisone 60 mg to healthy individuals and monitor them for the next  $6-6\frac{1}{2}$  hours after the administration of the drug. It is unlikely that any harmful side effects will occur with a single exposure to

glucocorticoids. Prednisone has a half-life of 18-36 hours; thus, we will instruct all the participants to contact us if they experience any discomfort within the next 72 hours after the study conclusion.

# 8.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

The proposed study is low risk. These studies do not fall into the traditional Phase I, II, or III clinical trial concepts. Nevertheless it is important to monitor the data obtained and subject safety. Monitoring should be commensurate with the risks, which are small. The principal investigator proposes to review the data weekly and adverse events if they occur. During the conduct of the study, any serious adverse event will be reported to the IRB within 7 days of the PI's notification of the event. Should the risk-benefit ratio of the study change the principal investigator will make alterations to the procedures of the study and submit them to the IRB.

# 9.0 Study Withdrawal/Discontinuation

Withdrawal of participants from any part or the whole study is under the discretion of the PI and will be done if:

- Performing a specific study procedure may be harmful for the participant or he/she cannot tolerate the procedure.
- The participant does not meet the study requirements
- The study is stopped
- Participant is not willing to continue the study

Participants who may not tolerate the OGTT may continue in the study to assess GC efficacy but not GC metabolic toxicity. The study team will explain to the participant why he/she is taken out from specific procedures or from the whole study.

#### 10.0 Statistical Considerations

Although this is a pilot study that will provide preliminary information of the effect size and variability of our outcomes (clinical and gene expression changes), we have 85% power to detect a minimum fold change of 2.5 for a total number of 20,000 tested genes with the top 100 being prognostic with a FDR of 0.1 using exact test, assuming a minimum average read counts of 10 for prognostic genes, a maximum dispersion of 0.5, and a ratio of the geometric mean of normalization factor of 1. The main analysis of the gene expression data will be carried out by Dr. Yan Guo (VANGARD), who will perform the following procedures:

- Detect genes that on average change expression levels due to GC treatment: we will normalized gene expression data. We will use the  $log_2$  fold change in expression as a measure of response, and perform multiple linear regression controlling for potential covariates (batch, age, and BMI) with a FDR < 0.1.
- Identify a set of genes with expression patterns are predictive of GC response: to test the association between changes in our clinical outcomes (lymphocyte counts and metabolic indexes) and log<sub>2</sub> fold change for each gene, we will perform linear regression analysis using a FDR of 0.1. We will stratify our analysis by sex. To control for the effect of estrogens levels in GC response among females, we will register the day of the menstrual cycle that the study visit occurred and include it as a covariate. For women

who are using a hormonal birth control method, we will also include the type of hormone birth control method (systemic or local), and active ingredient (progesterone with and without estrogen) as covariates.

• Select a list of candidate of regulatory variants that are likely to explain the observed variability in gene expression patterns: using public available eQTL datasets (GTEx, seeQTL, NCBI eQTL Browser, Genevar, SCAN, ExSNP, etc), we will query genes that their gene expression profile are predictive of GC response to identify a candidate list of variants for genome interrogation. We will select variants that: (a) have shown to be significantly associated with the expression of the respective gene (P<5x10<sup>-4</sup>), (b) are located within 1 megabase on either site of the gene's transcriptional start site, and (c) have MAF >0.10. We will combined genome information and the gene expression data using a Bayes factor calculation<sup>27</sup> to identify which variants do affect gene expression profile with GC administration with and without OGTT.

Additionally, to determine which mechanisms are shared between in *in vivo* and *in vitro* GC exposure, we plan to culture PBMCs with GC in normoglycemic and hyperglycemic media. PBMCs will be isolate from blood samples collected at screening visit and culture for 4 hours with GC in a normoglycemic and hyperglycemic media to simulate the effect of OGTT and measure changes in gene expression. By comparing gene expression profiles from *in vivo* and *in vitro* administration of GC on PBMCs from the same individual, we can identify which mechanisms are shared in both conditions. This will largely improve our ability to perform clinical studies in the future that involve GC exposure by reducing the risk and costs related to drug exposure for specific mechanisms that are shared in *in vitro* and *in vivo* response.

# 11.0 Privacy/Confidentiality Issues

Confidentiality and ethical considerations will be addressed as follows. All identifying documents, data, and specimens collected as a result of this study will be retained by the investigator. The information collected will be stored in a secure, password-protected database. All samples collected will be labeled with a unique code. Access to this material will be available only to the research investigator and/or her research staff. If results of this study are to be published, only code numbers will be used for identification purposes. Participants will not be identified by name.

#### 12.0 Follow-up and Record Retention

For this pilot study, we expect to finish participant enrollment within 2 years. However, we expect that the sequencing process, genome interrogation, and data analysis will be completed within 3 years. Research data that results from this study will be archive for unknown length of time.

#### Reference List

- 1. Fardet L, Petersen I, Nazareth I. Prevalence of long-term oral glucocorticoid prescriptions in the UK over the past 20 years. Rheumatology (Oxford) 2011;50(11):1982-1990.
- 2. Barnes PJ, Adcock IM. Glucocorticoid resistance in inflammatory diseases. Lancet 2009;373(9678):1905-1917.
- 3. Overman RA, Yeh JY, Deal CL. Prevalence of oral glucocorticoid usage in the United States: A general population perspective. Arthritis Care Res (Hoboken ) 2012.
- 4. Leung DY, Bloom JW. Update on glucocorticoid action and resistance. J Allergy Clin Immunol 2003;111(1):3-22.
- 5. Chan MT, Leung DY, Szefler SJ, Spahn JD. Difficult-to-control asthma: clinical characteristics of steroid-insensitive asthma. J Allergy Clin Immunol 1998;101(5):594-601.
- 6. Faubion WA, Jr., Loftus EV, Jr., Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of corticosteroid therapy for inflammatory bowel disease: a population-based study. Gastroenterology 2001;121(2):255-260.
- 7. van SD, Valkema R, Dijkmans BA et al. Prednisone treatment of elderly-onset rheumatoid arthritis. Disease activity and bone mass in comparison with chloroquine treatment. Arthritis Rheum 1995;38(3):334-342.
- 8. Barnes PJ, Jonsson B, Klim JB. The costs of asthma. Eur Respir J 1996;9(4):636-642.
- 9. Mazzantini M, Torre C, Miccoli M et al. Adverse events during longterm low-dose glucocorticoid treatment of polymyalgia rheumatica: a retrospective study. J Rheumatol 2012;39(3):552-557.
- 10. Saag KG, Koehnke R, Caldwell JR et al. Low dose long-term corticosteroid therapy in rheumatoid arthritis: an analysis of serious adverse events. Am J Med 1994;96(2):115-123.
- 11. Proven A, Gabriel SE, Orces C, O'Fallon WM, Hunder GG. Glucocorticoid therapy in giant cell arteritis: duration and adverse outcomes. Arthritis Rheum 2003;49(5):703-708.
- 12. Tantisira KG, Lasky-Su J, Harada M et al. Genomewide association between GLCCI1 and response to glucocorticoid therapy in asthma. N Engl J Med 2011;365(13):1173-1183.

- 13. Tantisira KG, Damask A, Szefler SJ et al. Genome-wide association identifies the T gene as a novel asthma pharmacogenetic locus. Am J Respir Crit Care Med 2012;185(12):1286-1291.
- 14. Qiu W, Rogers AJ, Damask A et al. Pharmacogenomics: novel loci identification via integrating gene differential analysis and eQTL analysis. Hum Mol Genet 2014;23(18):5017-5024.
- 15. McGeachie MJ, Wu AC, Chang HH, Lima JJ, Peters SP, Tantisira KG. Predicting inhaled corticosteroid response in asthma with two associated SNPs. Pharmacogenomics J 2012.
- 16. Mager DE, Lin SX, Blum RA, Lates CD, Jusko WJ. Dose equivalency evaluation of major corticosteroids: pharmacokinetics and cell trafficking and cortisol dynamics. J Clin Pharmacol 2003;43(11):1216-1227.
- 17. Magee MH, Blum RA, Lates CD, Jusko WJ. Pharmacokinetic/pharmacodynamic model for prednisolone inhibition of whole blood lymphocyte proliferation. Br J Clin Pharmacol 2002;53(5):474-484.
- 18. Fauci AS. Mechanisms of corticosteroid action on lymphocyte subpopulations. I. Redistribution of circulating T and b lymphocytes to the bone marrow. Immunology 1975;28(4):669-680.
- 19. Dale DC, Fauci AS, Guerry D, IV, Wolff SM. Comparison of agents producing a neutrophilic leukocytosis in man. Hydrocortisone, prednisone, endotoxin, and etiocholanolone. J Clin Invest 1975;56(4):808-813.
- 20. Fardet L, Flahault A, Kettaneh A et al. Corticosteroid-induced clinical adverse events: frequency, risk factors and patient's opinion. Br J Dermatol 2007;157(1):142-148.
- 21. Fardet L, Kassar A, Cabane J, Flahault A. Corticosteroid-induced adverse events in adults: frequency, screening and prevention. Drug Saf 2007;30(10):861-881.
- 22. Gurwitz JH, Bohn RL, Glynn RJ, Monane M, Mogun H, Avorn J. Glucocorticoids and the risk for initiation of hypoglycemic therapy. Arch Intern Med 1994;154(1):97-101.
- 23. Nicolae DL, Gamazon E, Zhang W, Duan S, Dolan ME, Cox NJ. Trait-associated SNPs are more likely to be eQTLs: annotation to enhance discovery from GWAS. PLoS Genet 2010;6(4):e1000888.
- 24. Albert FW, Kruglyak L. The role of regulatory variation in complex traits and disease. Nat Rev Genet 2015;16(4):197-212.
- 25. Li H, Pouladi N, Achour I et al. eQTL networks unveil enriched mRNA master integrators downstream of complex disease-associated SNPs. J Biomed Inform 2015;58:226-234.

- 26. Luca F, Maranville JC, Richards AL, Witonsky DB, Stephens M, Di RA. Genetic, functional and molecular features of glucocorticoid receptor binding. PLoS One 2013;8(4):e61654.
- 27. Maranville JC, Luca F, Richards AL et al. Interactions between glucocorticoid treatment and cis-regulatory polymorphisms contribute to cellular response phenotypes. PLoS Genet 2011;7(7):e1002162.
- 28. Fauci AS, Dale DC, Balow JE. Glucocorticosteroid therapy: mechanisms of action and clinical considerations. Ann Intern Med 1976;84(3):304-315.
- 29. Fauci AS, Dale DC. Alternate-day prednisone therapy and human lymphocyte subpopulations. J Clin Invest 1975;55(1):22-32.
- 30. Cupps TR, Fauci AS. Corticosteroid-mediated immunoregulation in man. Immunol Rev 1982;65:133-155.
- 31. Saavedra-Delgado AM, Mathews KP, Pan PM, Kay DR, Muilenberg ML. Doseresponse studies of the suppression of whole blood histamine and basophil counts by prednisone. J Allergy Clin Immunol 1980;66(6):464-471.
- 32. Barth J, Damoiseaux M, Mollmann H, Brandis KH, Hochhaus G, Derendorf H. Pharmacokinetics and pharmacodynamics of prednisolone after intravenous and oral administration. Int J Clin Pharmacol Ther Toxicol 1992;30(9):317-324.
- 33. Chakraborty A, Blum RA, Cutler DL, Jusko WJ. Pharmacoimmunodynamic interactions of interleukin-10 and prednisone in healthy volunteers. Clin Pharmacol Ther 1999;65(3):304-318.
- 34. Mishler JM, Emerson PM. Development of Neutrophilia by serially increasing doses of dexamethasone. Br J Haematol 1977;36(2):249-257.
- 35. Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. Clin Pharmacokinet 2005;44(1):61-98.
- 36. Shoenfeld Y, Gurewich Y, Gallant LA, Pinkhas J. Prednisone-induced leukocytosis. Influence of dosage, method and duration of administration on the degree of leukocytosis. Am J Med 1981;71(5):773-778.
- 37. Serra-Bonett N, Al SS, Rodriguez MA. Effect of low-dose prednisone on leukocyte counts and subpopulations in patients with rheumatoid arthritis. J Clin Rheumatol 2009;15(3):148-149.
- 38. Donihi AC, Raval D, Saul M, Korytkowski MT, DeVita MA. Prevalence and predictors of corticosteroid-related hyperglycemia in hospitalized patients. Endocr Pract 2006;12(4):358-362.

- 39. Kwon S, Hermayer KL. Glucocorticoid-induced hyperglycemia. Am J Med Sci 2013;345(4):274-277.
- 40. Clore JN, Thurby-Hay L. Glucocorticoid-induced hyperglycemia. Endocr Pract 2009;15(5):469-474.
- 41. Bergman RN, Finegood DT, Kahn SE. The evolution of beta-cell dysfunction and insulin resistance in type 2 diabetes. Eur J Clin Invest 2002;32 Suppl 3:35-45.
- 42. DeFronzo RA. Pathogenesis of type 2 diabetes mellitus. Med Clin North Am 2004;88(4):787-835, ix.
- 43. Yuen KC, Chong LE, Riddle MC. Influence of glucocorticoids and growth hormone on insulin sensitivity in humans. Diabet Med 2013;30(6):651-663.
- 44. van Raalte DH, Nofrate V, Bunck MC et al. Acute and 2-week exposure to prednisolone impair different aspects of beta-cell function in healthy men. Eur J Endocrinol 2010;162(4):729-735.
- 45. Hollingdal M, Juhl CB, Dall R et al. Glucocorticoid induced insulin resistance impairs basal but not glucose entrained high-frequency insulin pulsatility in humans. Diabetologia 2002;45(1):49-55.
- 46. Kauh E, Mixson L, Malice MP et al. Prednisone affects inflammation, glucose tolerance, and bone turnover within hours of treatment in healthy individuals. Eur J Endocrinol 2012;166(3):459-467.
- 47. Abdelmannan D, Tahboub R, Genuth S, Ismail-Beigi F. Effect of dexamethasone on oral glucose tolerance in healthy adults. Endocr Pract 2010;16(5):770-777.
- 48. Taheri N, Aminorroaya A, Ismail-Beigi F, Amini M. Effect of dexamethasone on glucose homeostasis in normal and prediabetic subjects with a first-degree relative with type 2 diabetes mellitus. Endocr Pract 2012;18(6):855-863.
- 49. Plat L, Byrne MM, Sturis J et al. Effects of morning cortisol elevation on insulin secretion and glucose regulation in humans. Am J Physiol 1996;270(1 Pt 1):E36-E42.
- 50. Larsson H, Ahren B. Insulin resistant subjects lack islet adaptation to short-term dexamethasone-induced reduction in insulin sensitivity. Diabetologia 1999;42(8):936-943.
- 51. Wajngot A, Giacca A, Grill V, Vranic M, Efendic S. The diabetogenic effects of glucocorticoids are more pronounced in low- than in high-insulin responders. Proc Natl Acad Sci U S A 1992;89(13):6035-6039.
- 52. Henriksen JE, Alford F, Ward GM, Beck-Nielsen H. Risk and mechanism of dexamethasone-induced deterioration of glucose tolerance in non-diabetic first-degree relatives of NIDDM patients. Diabetologia 1997;40(12):1439-1448.

- 53. Grill V, Pigon J, Hartling SG, Binder C, Efendic S. Effects of dexamethasone on glucose-induced insulin and proinsulin release in low and high insulin responders. Metabolism 1990;39(3):251-258.
- 54. Iwamoto T, Kagawa Y, Naito Y, Kuzuhara S, Kojima M. Steroid-induced diabetes mellitus and related risk factors in patients with neurologic diseases. Pharmacotherapy 2004;24(4):508-514.
- 55. Tornatore KM, Biocevich DM, Reed K, Tousley K, Singh JP, Venuto RC. Methylprednisolone pharmacokinetics, cortisol response, and adverse effects in black and white renal transplant recipients. Transplantation 1995;59(5):729-736.
- 56. Fennell RS, Van DJ, Riley WJ. Steroid-induced diabetes in pediatric renal transplant recipients. Int J Pediatr Nephrol 1983;4(2):103-107.
- 57. van Rossum EF, Koper JW, Huizenga NA et al. A polymorphism in the glucocorticoid receptor gene, which decreases sensitivity to glucocorticoids in vivo, is associated with low insulin and cholesterol levels. Diabetes 2002;51(10):3128-3134.
- 58. Syed AA, Halpin CG, Irving JA et al. A common intron 2 polymorphism of the glucocorticoid receptor gene is associated with insulin resistance in men. Clin Endocrinol (Oxf) 2008;68(6):879-884.
- 59. van Raalte DH, van LN, Simonis-Bik AM et al. Glucocorticoid receptor gene polymorphisms are associated with reduced first-phase glucose-stimulated insulin secretion and disposition index in women, but not in men. Diabet Med 2012;29(8):e211-e216.
- 60. Trementino L, Appolloni G, Concettoni C, Cardinaletti M, Boscaro M, Arnaldi G. Association of glucocorticoid receptor polymorphism A3669G with decreased risk of developing diabetes in patients with Cushing's syndrome. Eur J Endocrinol 2012;166(1):35-42.
- 61. Giordano R, Marzotti S, Berardelli R et al. BCII polymorphism of the glucocorticoid receptor gene is associated with increased obesity, impaired glucose metabolism and dyslipidaemia in patients with Addison's disease. Clin Endocrinol (Oxf) 2012;77(6):863-870.
- 62. Di Blasio AM, van Rossum EF, Maestrini S et al. The relation between two polymorphisms in the glucocorticoid receptor gene and body mass index, blood pressure and cholesterol in obese patients. Clin Endocrinol (Oxf) 2003;59(1):68-74.
- 63. Huizenga NA, Koper JW, de LP et al. Interperson variability but intraperson stability of baseline plasma cortisol concentrations, and its relation to feedback sensitivity of the hypothalamo-pituitary-adrenal axis to a low dose of dexamethasone in elderly individuals. J Clin Endocrinol Metab 1998;83(1):47-54.

- 64. Dobson MG, Redfern CP, Unwin N, Weaver JU. The N363S polymorphism of the glucocorticoid receptor: potential contribution to central obesity in men and lack of association with other risk factors for coronary heart disease and diabetes mellitus. J Clin Endocrinol Metab 2001;86(5):2270-2274.
- 65. Goracy I, Goracy J, Safranow K, Skonieczna-Zydecka K, Ciechanowicz A. Association of glucocorticoid receptor gene NR3C1 genetic variants with angiographically documented coronary artery disease and its risk factors. Arch Med Res 2013;44(1):27-33.
- 66. Grundberg E, Adoue V, Kwan T et al. Global analysis of the impact of environmental perturbation on cis-regulation of gene expression. PLoS Genet 2011;7(1):e1001279.
- 67. Maranville JC, Baxter SS, Torres JM, Di RA. Inter-ethnic differences in lymphocyte sensitivity to glucocorticoids reflect variation in transcriptional response. Pharmacogenomics J 2013;13(2):121-129.
- 68. Gordon K, Clouaire T, Bao XX et al. Immortality, but not oncogenic transformation, of primary human cells leads to epigenetic reprogramming of DNA methylation and gene expression. Nucleic Acids Res 2014;42(6):3529-3541.
- 69. Lorsch JR, Collins FS, Lippincott-Schwartz J. Cell Biology. Fixing problems with cell lines. Science 2014;346(6216):1452-1453.
- 70. Zaitseva M, Vollenhoven BJ, Rogers PA. In vitro culture significantly alters gene expression profiles and reduces differences between myometrial and fibroid smooth muscle cells. Mol Hum Reprod 2006;12(3):187-207.
- 71. Olnes MJ, Kotliarov Y, Biancotto A et al. Effects of Systemically Administered Hydrocortisone on the Human Immunome. Sci Rep 2016;6:23002.
- 72. Dalla MC, Campioni M, Polonsky KS et al. Two-hour seven-sample oral glucose tolerance test and meal protocol: minimal model assessment of beta-cell responsivity and insulin sensitivity in nondiabetic individuals. Diabetes 2005;54(11):3265-3273.
- 73. Cobelli C, Toffolo GM, Dalla MC et al. Assessment of beta-cell function in humans, simultaneously with insulin sensitivity and hepatic extraction, from intravenous and oral glucose tests. Am J Physiol Endocrinol Metab 2007;293(1):E1-E15.